CLINICAL TRIAL: NCT02227212
Title: A Multi-Center,Open-Label, Single-Arm, Multiple Dose Study With HOE901-U300 to Assess The Ease of Use And Safety of a New U300 Pen Injector in Insulin-Naïve Patients With T2DM
Brief Title: Ease of Use and Safety of the New U300 Pen Injector in Insulin-Naïve Patients With T2DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDY14065; 2014-001253-16; U1111-1155-7309 (Other: UTN)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin glargine U300 (Experimental): Once daily subcutaneous injection for 4 weeks
  Interventions: Drug: Insulin glargine U300 (new formulation of insulin glargine) HOE901

INTERVENTIONS:
Drug: Insulin glargine U300 (new formulation of insulin glargine) HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To demonstrate the ease of use of the U300 pen injector in pen-naïve and insulin-naïve type 2 diabetes mellitus (T2DM) patients in a 4-week once-daily dosing regimen with HOE901-U300.

Secondary Objectives:

To assess in a 4-week once-daily dosing regimen with HOE901-U300 in pen-naïve and insulin-naïve T2DM patients.

The safety and usability of the U300 pen injector. The glycemic control with the U300 pen injector. The safety of HOE901-U300.

DETAILED DESCRIPTION:
The total study duration for a participants can be approximately up to 10 weeks.

ELIGIBILITY:
Inclusion criteria:

* Patients with T2DM inadequately controlled with non-insulin, non-injectable anti-hyperglycemic drug(s) and for whom the Investigator/treating physicians has decided that basal insulin is appropriate.
* Signed written informed consent.

Exclusion criteria:

* Glycated hemoglobin A1c (HbA1c) <7.0% (<53 mmol/mol) or >11% (97 mmol/mol) at screening.
* Age <18 years at the time of screening.
* Body Mass Index (BMI) >40 kg/m2.
* Diabetes other than T2DM.
* History of T2DM for less than 1 year before screening.
* Less than 6 months anti-hyperglycemic treatment before screening.
* Initiation of new glucose-lowering medications and/or weight loss drug in the last 3 months before screening visit.
* Previous treatment with Glucagon Like Peptide-1 (GLP-1) agonist.
* Patients receiving only non-insulin anti-hyperglycemic drugs not approved for combination with insulin according to local labeling/local treatment guidelines and/or sulfonylurea or glinides.
* Current or previous insulin use except for a maximum of 8 consecutive days and a total of 14 days (eg, acute illness, surgery) during the last year prior to screening.
* Any contraindication to insulin glargine (Lantus) according to the National Product labeling or any excipients.
* Any contraindication to the mandatory background non-insulin anti-hyperglycemic medication according to the respective National Product labeling.
* Latest eye examination by an ophthalmologist >12 months prior to inclusion.
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months.
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment or injectable drugs) during the study period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Ease-of-use / ease of learning questionnaire | Day 1, Day 7 , 4-weeks

SECONDARY OUTCOMES:
Change in treatment satisfaction score (sum of items 1, 4, 5, 6, 7, and 8 from Diabetes Treatment Satisfaction Questionnaire [status]) from baseline to Week 4 | Baseline, week 4
Change in perception of hyper- and hypoglycemia score (items 2 and 3 from Diabetes Treatment Satisfaction Questionnaire [status]) from baseline to Week 4 | Baseline, week 4
Change in fasting plasma glucose (FPG) (mmol/L) from baseline to Week 4 | Baseline, week 4
Number of participants with Product Technical Complaints (PTC) | Baseline to week 4
Number of participants with adverse events and hypoglycemic events related to PTC | Baseline to week 4
Change in daily insulin dose (U and U/kg) from Day 1 to Week 4 (patient diary) | Baseline, week 4
Number of participants with adverse events | screening to week 6
Incidence and frequency of hypoglycemia episodes. Hypoglycemia will be analyzed by hypoglycemia categories as defined by American Diabetes Association | screening to week 6
Potentially clinically significant changes in laboratory evaluations, vital signs, electrocardiogram (ECG) | screening, baseline, week 4
Number of participants with site injection site reactions / hypersensitivity reactions | baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (7):
- Germany (7):
  - Investigational Site Number 276011, Augsburg
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276009, Essen
  - Investigational Site Number 276002, Hamburg
  - Investigational Site Number 276001, Münster
  - Investigational Site Number 276007, Potsdam
  - Investigational Site Number 276004, Wangen

REFERENCES:
- [Derived] Pohlmeier H, Berard L, Brulle-Wohlhueter C, Wu J, Dahmen R, Nowotny I, Klonoff D. Ease of Use of the Insulin Glargine 300 U/mL Pen Injector in Insulin-Naive People With Type 2 Diabetes. J Diabetes Sci Technol. 2017 Mar;11(2):263-269. doi: 10.1177/1932296816668877. Epub 2016 Sep 25. PMID 27664062